CLINICAL TRIAL: NCT00029198
Title: Preterm Infants' Weight Gain Following Massage Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Tiffany Field, Director, Touch Research Institute, University of Miami
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: R01AT000370-01 (NIH); R01AT000370-01 (NIH); R01AT000370 (NIH)
Record Dates: First submitted 2002-01-09; First posted 2002-01-10 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Premature Birth
Keywords: Massage Therapy; Preterm Infants; Weight Gain; Vagal Tone; IGF-1; Oxytocin; Brazelton
MeSH Terms: conditions — Premature Birth; Weight Gain | interventions — Massage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 15 minute massage tid
  Interventions: Procedure: massage
- 2 (Sham Comparator): non-massage touch
  Interventions: Procedure: Sham massage

INTERVENTIONS:
Procedure: massage — 15 massage given tid
  Arms: 1
Procedure: Sham massage — non-massage touch
  Arms: 2

SUMMARY:
The specific aims of this study are: 1) to replicate the data that following ten days of massage therapy, preterm infants show greater daily weight gain and are discharged from the hospital earlier than the controls, thus demonstrating the cost-effectiveness of the intervention; 2) to test a model on two potential underlying mechanisms for weight gain including a) enhanced vagal activity leading to greater gastric motility, higher levels of insulin, IGF-1, and oxytocin and lower cortisol levels in the massage versus the control infants at the end of the study; and/or b) increased physical activity and its associated increase in heart rate oxygen consumption and temperature leading to greater weight gain. These pathways (vagal activity and physical activity) will be tested by path analyses. Determining underlying mechanisms for the massage therapy/weight gain relationship is a critical process required by the neonatology community for massage therapy to be adopted as a standard neonatal intensive care unit.

DETAILED DESCRIPTION:
A number of studies have documented an average of 47% greater weight gain in preterm neonates following massage therapy. Our currently funded study suggests that massage therapy increases vagal activity, oxytocin, and IGF-1. In the proposed continuation of this study preemies would be provided daily massages three times a day for 10 days, as in our previously successful protocol. To determine potential mechanisms that may underlie the massage therapy/weight gain relationship we will continue to assess vagal activity and assay insulin, oxytocin, IGF-1 and cortisol as well as gastric motility. We have added an alternative potential pathway for the massage therapy/weight gain relationship. In this expanded model, activity level and the related measures of heart rate, oxygen consumption (based on a formula calculated from heart rate) and temperature mediate the effects of massage therapy on weight gain. A larger sample will be recruited so that we can have the power needed to test our model of the potential mechanisms underlying the weight gain from preterm infant massage. For the current application, 120 preterm infants with common medical complications of prematurity, who are medically stable and residing in the intermediate care ("grower") nursery, will be assigned to groups based on a random stratification on the following variables: gender, gestational age, birthweight, days in the NICU, and study entry weight. One hundred twenty infants will be randomly assigned to one of two groups: 1) ten days of massage therapy (n=60), or 2) standard treatment (n=60). Within-subjects and between-groups analyses will focus on physiological (heart rate, vagal tone, gastric motility, and temperature), biochemical (insulin, oxytocin, IGF-1 and cortisol) and behavioral variables (activity level).

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 28 and 32 weeks
* Birthweight between 800 and 1,400 grams
* Birthweight, length, and head circumference appropriate for gestational age
* Scores on the Obstetric/Postnatal Complications scales are each below 80
* NICU stay between 15 and 60 days
* Current weight between 1,000 and 1,500 grams
* Current daily intake is between 120 and 160 calories

Exclusion Criteria:

* Genetic anomalies, congenital heart malformations, and/or central nervous system dysfunction
* HIV infection
* History of maternal alcohol or illicit drug use
* Syphilis
* Hepatitis B
* Require surgery

Ages: 28 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 139 (Actual)
Dates: Start 2003-04; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
weight gain | post-massage

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany M Field, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami School of Medicine, Miami, Florida, United States

REFERENCES:
- [Derived] Field T, Diego M, Hernandez-Reif M, Dieter JN, Kumar AM, Schanberg S, Kuhn C. Insulin and insulin-like growth factor-1 increased in preterm neonates following massage therapy. J Dev Behav Pediatr. 2008 Dec;29(6):463-6. doi: 10.1097/DBP.0b013e3181856d3b. PMID 18714203
- See also: Touch Research Institutes — http://www.miami.edu/touch-research